CLINICAL TRIAL: NCT05669326
Title: Evaluation of the Contribution of NODDI Protocol Tractography in Brain Tumor Surgery
Acronym: NODDI-TRACT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No recrutment
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-A02074-37
Record Dates: First submitted 2022-12-20; First posted 2022-12-30 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Malignant Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NODDI TRACT (Experimental): * Diffusion MRI (tractography) Tractography is performed on the basis of a diffusion MRI sequence which, after computer processing, will result in a map of the apparent diffusion coefficient and a diffusion tensor beam reconstruction (DTI tractography) performed with the Sisyphus software.
  * Multi-shell diffusion MRI (NODDI-tract)
  Interventions: Other: NODDI TRACT

INTERVENTIONS:
Other: NODDI TRACT — Compared to their usual management, the participation of the patient in this study implies an additional visit during which an MRI examination without contrast injection will be performed, lasting approximately 40 minutes (including installation and deinstallation).
  The operative time, surgical procedures and postoperative follow-up are not modified in this study.

SUMMARY:
The objective of this study is to evaluate to what extent the capacity of the NODDI model can allow, in case of Malignant brain tumor patients with vasogenic edema, the elaboration of a reliable cerebral functional mapping in accordance with the data of direct electrical stimulation (DES) which is today the reference tool.

the patient's participation in this study implies an additional visit during which an MRI examination without injection of contrast medium will be performed, lasting approximately 40 minutes (including installation and de-installation).

DETAILED DESCRIPTION:
This is a single-center, prospective, open-label study of neurosurgical patients.

Compared to their usual management, the participation of the patient in this study implies an additional visit during which an MRI examination without injection of contrast product will be performed, lasting approximately 40 minutes (including installation and de-installation).

The operative time, surgical procedures and postoperative follow-up are not modified in this study

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older,
* Patient who has read and signed the consent form for participation in the study
* Patient requiring surgery for a malignant brain tumor with vasogenic edema
* Patient with an estimated life expectancy of more than 3 months.

Exclusion Criteria:

* Patient under legal protection, guardianship or trusteeship
* Patient not affiliated to the French social security system
* Contraindication to MRI (patient with a pacemaker or cardiac defibrillator, implanted equipment activated by an electrical, magnetic or mechanical system, patient with hemostatic clips on intracerebral aneurysms or with orthopedic implants, claustrophobic patient)
* Psychiatric history
* Refusal to be informed of an abnormality detected during the MRI
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Response to electrical stimulation | Hour 24
  Response to electrical stimulation, which determines the presence or absence of an essential bundle, is the primary end point.
  The ability of the NODDI-tract method to reconstruct essential bundles in vasogenic edema will be assessed by estimating the correspondence between the response to intraoperative direct electrical stimulation (DES) and the presence of an MRI reconstructed bundle.
  Based on the response to electrical stimulation, the NODDI-tract data will be classified into one of four groups:
  * True positive = response to stimulation and presence of an MRI beam
  * True negative = no response to stimulation and no beam on MRI
  * False positive = no response to stimulation and presence of a beam on MRI
  * False-negative = response to stimulation and absence of beam in MRI. The distance between the reconstructed beam and the stimulation point (whether or not the stimulation was effective) will also be measured.

SECONDARY OUTCOMES:
Number of reconstructed fibers | Hour 24
  Reconstructions obtained using the NODDI protocol or tractography will be compared on the total number of fibers reconstructed by both methods.
  The comparison will be made on the total number of reconstructed fibers and on the number of reconstructed fibers crossing the edema.
Average distance to a reference atlas | Hour 24
  The comparison is based on the evaluation of the average distance between the skeleton of the NODDI-tract reconstructed beams and that of the JHU tractography atlas [20]. The distance will be calculated by projecting the reconstructed skeleton onto the atlas skeleton, and as a function of the length traveled on the parameterized curve representing the skeleton. This function will be averaged over the entire length of the skeleton. An average distance of less than 1cm will be considered as a match criterion.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de l'Union, Saint-Jean, France

IPD SHARING:
Plan to Share IPD: No